CLINICAL TRIAL: NCT06688409
Title: Comparing Home Blood Pressure Measurements from Devices with and Without Evidence of Validation to Ambulatory Blood Pressure Monitoring: the VALID-HomeBP Study
Brief Title: Accuracy Testing of Validated and Non-validated Home BP Devices Sold on the Online Market.
Acronym: VALID-HomeBP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Responsible Party: Principal Investigator, Remi Goupil, MD MSc, Principal investigator, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: VALID-HomeBP
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Hypertension
Keywords: hypertension; blood pressure measurement; blood pressure; blood pressure device validation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Validate home BP device (Active Comparator): BP measured with a validated home BP device
  Interventions: Diagnostic Test: awake ABPM
- Non-validated home BP device #1 (Active Comparator): BP measured with the first non-validated home BP device
  Interventions: Diagnostic Test: awake ABPM
- Non-validated home BP device #2 (Active Comparator): BP measured with the second non-validated home BP device
  Interventions: Diagnostic Test: awake ABPM
- Non-validated home BP device #3 (Active Comparator): BP measured with the third non-validated home BP device
  Interventions: Diagnostic Test: awake ABPM

INTERVENTIONS:
Diagnostic Test: awake ABPM — Comparison of a BP measured with the home BP devices and the average awake ABPM performed immediately after

SUMMARY:
This study aims to assess whether validated and non-validated blood pressure measuring devices sold on the online market are accurate in regards to the mean awake BP from ambulatory blood pressure monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged > 18 years scheduled to undergo an ABPM

Exclusion Criteria:

* Upper arm size outside of cuff range of selected devices (<22 cm or >42 cm)
* Night shift workers
* Permanent atrial fibrillation
* Known severe aortic stenosis
* Contraindication to measure BP on the non-dominant arm
* Ongoing pregnancy
* Inability or unwillingness to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Mean difference in systolic BP | At enrollment (time 0)
  Mean difference in systolic BP between the home BP device and the awake ABPM

SECONDARY OUTCOMES:
Mean difference in diastolic BP | At enrollment (time 0)
  Mean difference in diastolic BP between the home BP device and the awake ABPM
Mean difference in systolic BP from validated device | At enrollment (time 0)
  Mean difference in systolic BP between the non-validated home BP device and the validated home BP device
Mean difference in diastolic BP from validated device | At enrollment (time 0)
  Mean difference in diastolic BP between the non-validated home BP device and the validated home BP device

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Sacré-Coeur de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided